CLINICAL TRIAL: NCT06274307
Title: Efficacy of Transversus Abdominis Plane Block in an Insufflated Abdomen
Brief Title: Efficacy of Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justin Hruska (Other)
Responsible Party: Sponsor-Investigator, Justin Hruska, Principal Investigator, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-21-10-4045
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia, Local
Keywords: Transversus abdominal-plane block; Pain managment; Ultrasound

STUDY DESIGN:
Intervention Model Description: The treatment group (Group 1) will have a transversus abdominis plane (TAP) block performed with an insufflated abdomen in the operating room. The control group (Group 2) will receive the traditionally performed standard of care TAP block performed in the post-anesthesia care unit
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be unaware of their grouping allotment. The outcomes assessor will be unaware of the patient grouping allotment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Transversus abdominis plane (TAP) block performed in operating room (Active Comparator): The treatment group will have a transversus abdominis plane (TAP) block performed prior to closing surgical port sites post-operatively in an insufflated abdomen in the operating room (OR). The local anesthetic used for the TAP block will be 30 to 40ml of Ropivacaine 0.375%, not to exceed a max dose of 3mg/kg of 0.375% divided equally bilaterally. Each study participant will receive standard post-operative pain medication orders of morphine 2mg q5mins times 4 doses followed by hydromorphone. 0.5mg q10mins times 4 doses.
  Interventions: Procedure: Transversus abdominis plane block
- Transversus abdominis plane (TAP) block performed in PACU (Active Comparator): The treatment group will have a transversus abdominis plane (TAP) block performed post-operatively after the patient has been transferred from the Operating Room to the Post Anesthesia Care Unit (PACU). The local anesthetic used for the TAP block will be 30 to 40ml of Ropivacaine 0.375%, not to exceed a max dose of 3mg/kg of 0.375% divided equally bilaterally. Each study participant will receive standard post-operative pain medication orders of morphine 2mg q5mins times 4 doses followed by hydromorphone. 0.5mg q10mins times 4 doses
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — A transversus abdominis plane block (TAP) block using a long-acting local anesthetic is used to manage pain during the intermediate (12-24hr) post-operative period following laparoscopic abdominal surgeries. Drug: The local anesthetic to be used in this specific intervention will be 30 to 40ml of Ropivacaine 0.375%, not to exceed a max dose of 3mg/kg of 0.375% and divided equally bilaterally.

SUMMARY:
This study aims to assess the efficacy of Transversus Abdominus Plane (TAP) blocks, a well-established anesthetic technique, to decrease the amount of post-operative pain in patients who undergo minimally invasive gynecologic surgeries. During minimally invasive gynecologic surgeries, the abdomen is inflated with pressurized air for visualization purposes and released at the end of the surgery. Traditionally, TAP blocks are performed by injecting long-acting local anesthetic agents under ultrasound guidance into the abdominal wall after abdominal surgery after the air has been emptied from the abdomen for additional anesthetic coverage post-operatively. This study proposes a novel approach: that performing TAP blocks while the abdomen is still insufflated will result in better post-operative pain outcomes as compared to the traditional method.

DETAILED DESCRIPTION:
Background

Every year 15 million laparoscopic procedures are performed globally, with 4,800,000 or 32% of procedures performed in the U.S. alone. This minimally invasive procedure is one of the most common surgical procedures in the United States. Approximately 350,000 or half of all bilateral tubal sterilizations are performed laparoscopically; almost two-thirds of the 600,000 hysterectomies are performed via laparoscopy. Laparoscopy is also commonly used for diagnostic purposes, and to perform other common procedures such as treatment for endometriosis and lysis of adhesions. During laparoscopic gynecologic surgeries, the surgical team will have the abdomen inflated with pressurized carbon dioxide for surgical visualization purposes which is then released at the end of the surgical procedure. For many laparoscopic procedures, a transversus abdominis plane block (TAP) block using a long-acting local anesthetic is used to manage pain performed outside the OR, more for logistical ease, traditionally this block is performed outside the operating room setting, in the post-operative period on a non- insufflated abdomen under ultrasound guidance.

Rationale for conducting the research. This study has two major aims; 1) to determine whether post-operative TAP blocks performed in an insufflated abdomen will result in more optimal postoperative pain control compared to TAP blocks performed in the traditional method in a non-insufflated abdomen and 2) to observe if performing the TAP block in a insufflated abdomen will be more clinically efficient to perform than the traditional method performed in a non-insufflated abdomen. The study hypothesis is that the study group receiving the TAP block the insufflated abdomen will have more optimal postoperative pain control, requiring less adjuvant pain medication as compared to the participants receiving the control intervention. Additionally, we hypothesize that the proceduralist will be able to perform a TAP block in less time with and with few attempts in the insufflated compared to the non- insufflated abdomen group due to better visualization of the anatomical planes from insufflation of the abdominal area. The results of this study may add additional clinically effective practice guidelines for both regional anesthesia and acute pain management relating to laparoscopic gynecological procedures. Furthermore, TAP blocks performed under insufflation may provide a viable method for decreasing opioid use and reducing potential opioid dependence in patients following surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female gynecological patients between 18 years and 85 years consented and scheduled for an obstetrics/gynecology laparoscopic procedure.
* Consent received to receive a TAP block.

Exclusion Criteria:

* Patients who are not proficient in the English language or cannot consent
* Patients who have an allergy to local anesthetics (amides)
* Patients with subcutaneous emphysema
* Patients whose surgical procedures require incisions above the umbilicus

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Time to perform TAP Block | Within 10 minutes of starting procedure.
  Time taken to successfully perform the TAP block. Defined as the time from initial placement of ultrasound probe on the skin to the completion of the block on the contralateral side.
TAP block attempts | Within 10 minutes of starting procedure.
  The number of attempts taken to sucessfully perform the TAP block.
Pain Score Visual Analog Scale (VAS) 0 Hours Post Surgery | 0 hours following TAP block]
  Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Pain Score Visual Analog Scale (VAS) 1 Hours Post Surgery | 1 hour following TAP block]
  Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Pain Score Visual Analog Scale (VAS) 2 Hours Post Surgery | 2 hours following TAP block]
  Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Pain Score Visual Analog Scale (VAS) 4 Hours Post Surgery | 4 hours following TAP block]
  Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Pain Score Visual Analog Scale (VAS) 24 Hours Post Surgery | 24 hours following TAP block]
  Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Postoperative Opioid Consumption | 24 hours post operative period
  Patient opioid consumption in the 24 hours post TAP block
Ease of performing TAP Block-anatomical plane visualization | Within 10 minutes of starting procedure
  The anatomical planes were clearly visualized and identified. Survey of operator - Likert Score
Ease of performing TAP Block-performance efficacy | Within 10 minutes of starting procedure
  The approach optimized the efficacy of the block. Survey of operator- Likert score
Patient satisfaction | 24-hours post operative period
  Patient satisfaction with analgesia score (0 to 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Hruska, MD, Principal Investigator — Wayne State University/Detroit Medical Center
Locations (2):
- United States (2):
  - Detroit Medical Center Detroit Receiving Hospital, Detroit, Michigan
  - Detroit Medical Center, Harper University Hospital, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No